CLINICAL TRIAL: NCT04728815
Title: Comprehensive Adaptive Multisite Prevention of University Student Suicide (CAMPUS) - Feasibility Sub-Study
Brief Title: CAMPUS - Feasibility Sub-Study
Acronym: CAMPUS-Feas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00104815; Pro00103346 (Other: Duke IRB); R01MH116062 (NIH); R01MH116052 (NIH); R01MH116050 (NIH); R01MH116061 (NIH)
Record Dates: First submitted 2021-01-25; First posted 2021-01-28 (Actual); Results first posted 2024-02-29 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Suicide
Keywords: Dialectical Behavior Therapy (DBT); Collaborative Assessment and Management of Suicide (CAMS); University Students
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of three treatments delivered via a hybrid model: (1) a suicide-focused treatment - Collaborative Assessment and Management of Suicidality (CAMS) for 4-8 weeks (n=35); (2) Treatment as Usual (TAU) for 4-8 weeks (n=15); or (3) Comprehensive Dialectical Behavior Therapy (DBT) for 16 weeks (n=35), which includes individual therapy, skills training, phone/text coaching for the clients, and peer consultation for the counselors.
  Sufficient responders to CAMS or TAU will discontinue services/be stepped down after 4-8 weeks. Non-responders to CAMS or TAU will be re-randomized to one of two higher intensity/dosage intervention options for an additional 8 weeks of treatment: (1) CAMS (either continued or administered for the first time) or (2) Comprehensive DBT.
  There is an 8th Arm/Group of Consented Study Counselors from each of the 4 sites.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- CAMS to Maintenance (Experimental): Subject assigned to CAMS for Phase 1. Subject is a Phase 1 CAMS Responder, thus placed into ongoing Maintenance/Monitoring.
  Interventions: Behavioral: CAMS - Phase 1
- CAMS to CAMS (Experimental): Subject assigned to CAMS for Phase 1. Subject is a Phase 1 CAMS Insufficient Responder, then assigned to Phase 2 CAMS.
  Interventions: Behavioral: CAMS - Phase 1; Behavioral: CAMS - Phase 2
- CAMS to DBT (Experimental): Subject assigned to CAMS for Phase 1. Subject is a Phase 1 CAMS Insufficient Responder, then assigned to Phase 2 DBT.
  Interventions: Behavioral: CAMS - Phase 1; Behavioral: DBT - Phase 2
- TAU to Maintenance (Experimental): Subject assigned to TAU for Phase 1. Subject is a Phase 1 TAU Responder, thus placed into ongoing Maintenance/Monitoring.
  Interventions: Behavioral: TAU - Phase 1
- TAU to CAMS (Experimental): Subject assigned to TAU for Phase 1. Subject is a Phase 1 TAU Insufficient Responder, then assigned to Phase 2 CAMS.
  Interventions: Behavioral: TAU - Phase 1; Behavioral: CAMS - Phase 2
- TAU to DBT (Experimental): Subject assigned to TAU for Phase 1. Subject is a Phase 1 TAU Insufficient Responder, then assigned to Phase 2 DBT.
  Interventions: Behavioral: TAU - Phase 1; Behavioral: DBT - Phase 2
- DBT Only (Experimental): Subject Assigned to DBT for Phase 1, continuing up to 16 weeks.
  Interventions: Behavioral: DBT - Phase 1 and 2
- Study Counselors (No Intervention): Consented Study Counselors from each of the 4 sites. Data collected regarding the Counselors is minimal and is maintained completely separately from the other 7 Student Participant Arms/Groups.

INTERVENTIONS:
Behavioral: TAU - Phase 1 — 4-8 weeks of TAU treatment
  Arms: TAU to CAMS; TAU to DBT; TAU to Maintenance
Behavioral: CAMS - Phase 1 — 4-8 weeks of CAMS treatment
  Arms: CAMS to CAMS; CAMS to DBT; CAMS to Maintenance
Behavioral: DBT - Phase 1 and 2 — up to 16 weeks of DBT treatment
  Arms: DBT Only
Behavioral: CAMS - Phase 2 — Up to 8 weeks of CAMS treatment
  Arms: CAMS to CAMS; TAU to CAMS
Behavioral: DBT - Phase 2 — Up to 8 weeks of DBT treatment
  Arms: CAMS to DBT; TAU to DBT

SUMMARY:
Suicide is the 2nd leading cause of death among college students and suicidal ideation and suicide-related behaviors are a frequent presenting problem at college counseling centers (CCCs), which are overburdened. Studies show that some students respond rapidly to treatment, whereas others require considerably more resources. Evidence-based adaptive treatment strategies (ATSs) are needed to address this heterogeneity in responsivity and complexity. ATSs individualize treatment via decision rules specifying how the type and intensity of an intervention can be sequenced based on risk factors, response, or compliance.

The purpose of this multisite study is to investigate the effectiveness of four adaptive treatment strategies (ATSs) to treat college students who report suicidal ideation when first seeking services at their college counseling center This multisite study will enroll moderately to severely suicidal college students in the "emerging adulthood" phase (ages 18-25) seeking services at CCCs. This Sequential Multi-Assignment Randomized Trial (SMART) will have two stages of intervention. In Stage 1, 700 participants from four CCCs will be randomized to 4-8 weeks of: 1) a suicide-focused treatment - Collaborative Assessment and Management of Suicidality (CAMS) or 2) Treatment as Usual (TAU). Sufficient responders to either intervention will discontinue services/be stepped down. Non-responders will be re-randomized to one of two Stage 2 higher intensity/dosage intervention options for an additional 4-16 weeks: 1) CAMS (either continued or administered for the first time) or 2) Comprehensive Dialectical Behavior Therapy (DBT), which includes individual therapy, skills group, and phone/text coaching for the clients and peer consultation for the counselors.

DETAILED DESCRIPTION:
We will enroll moderately to severely suicidal college students in the "emerging adulthood" phase (ages 18-25) seeking services at CCCs. Eighty-Five participants (N=85) from four CCCs will be randomized to one of three treatments delivered via a hybrid model: (1) a suicide-focused treatment - Collaborative Assessment and Management of Suicidality (CAMS) for 4-8 weeks (n=35); (2) Treatment as Usual (TAU) for 4-8 weeks (n=15); or (3) Comprehensive Dialectical Behavior Therapy (DBT) for 16 weeks (n=35), which includes individual therapy, skills training, phone/text coaching for the clients, and peer consultation for the counselors.

Sufficient responders to CAMS or TAU will discontinue services/be stepped down after 4-8 weeks. Non-responders to CAMS or TAU will be re-randomized to one of two higher intensity/dosage intervention options for an additional 8 weeks of treatment: (1) CAMS (either continued or administered for the first time) or (2) Comprehensive DBT.

For the feasibility study, we will also enroll 12 CCC counselors (3 per site) who will serve as study counselor participants and periodically complete measures focused on the experience of counselors working with suicidal college students.

ELIGIBILITY:
Inclusion Criteria:

1. Enrolled at the university;
2. Eligible to receive counseling services either in person or remotely at the campus CCC (e.g., some students who are living in specific states may not be eligible for therapeutic services).
3. 18 to 25 years of age;
4. Moderate to severe SI over the last two weeks indicated by a score of greater than or equal to 2 on the Counseling Center Assessment of Psychological Symptoms (CCAPS-34) question, "I have thoughts of ending my life" (range is 0 "not at all like me" to 4 "extremely like me"); and
5. Agree to video recording of all therapy and assessment sessions.

Exclusion Criteria:

1. Students who are deemed clinically inappropriate to receive services at the CCC by an intake counselor because of imminent risk, severe psychosis, or inability to remain enrolled in school (e.g., academic failure);
2. Students being unable to remain enrolled in their university long enough to go through the minimum number of sessions for Stage 1 (4 sessions);
3. Students who have received services at the CCC within the last three months (i.e., ATSs must be based on a new treatment episode).

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2022-10-15 (Actual); Study Completion 2022-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Compton, PhD, Principal Investigator — Duke University; Jacqueline Pistorello, PhD, Principal Investigator — University of Nevada at Reno (UNR); Shireen Rizvi, PhD, Principal Investigator — Rutgers University; John Seeley, PhD, Principal Investigator — University of Oregon
Locations (4):
- United States (4):
  - University of Nevada - Reno, Reno, Nevada
  - Rutgers University, New Brunswick, New Jersey
  - Duke University, Durham, North Carolina
  - University of Oregon, Eugene, Oregon

IPD SHARING:
Plan to Share IPD: Yes
We will participant de-identified data (linked only by GUID) with the National Institute of Mental Health Data Archive (NDA). The NDA is an informatics system and research data repository developed by the National Institutes of Health (NIH) to share research data. The NDA provides the infrastructure to store, search across, and analyze various types of data. In addition, The NDA provides longitudinal storage of a research participant's information generated by one or more research studies. In other words, the NDA is able to associate a single research participant's genomic, imaging, clinical assessment and other information even if the data were collected at different locations or through different studies. By doing so, the NDA gives researchers access to more data than they can collect on their own, making it easier and faster for researchers to gather, evaluate, and share research information from a variety of sources.
Supporting Information: Study Protocol, SAP
Time Frame: All subject data will be submitted for inclusion in the NDA, through the conclusion of data collection activities. Data is to be submitted cumulatively, every 6 months.
Access Criteria: The NIH will provide access to scientific investigators for research purposes. Qualified researchers who have completed a Data Use Certification and received approval from the NDA Data Access Committee (DAC) may be approved to access broadly shared data. A separate request process exists for access to data in federated sources. Additionally, the DAC and support staff at NIH have access to NDA shared data.
URL: https://nda.nih.gov/nda/about-us.html

REFERENCES:
- [Derived] Kassing F, Seeley JR, Rizvi SL, Compton SN, Sinclair J, Oshin LA, Blalock K, Jobes DA, Crumlish J, Stadelman S, Gozenman-Sapin F, Snyderman T, Ruork AK, Fry CM, Gallop RJ, Goodrich J, Pistorello J. Assessing the implementation of suicide-focused treatments delivered in hybrid telemental health format in a real-world setting. Psychother Res. 2025 Sep;35(7):1198-1212. doi: 10.1080/10503307.2024.2415104. Epub 2024 Oct 22. PMID 39439041

RESULTS

PARTICIPANT FLOW:
Recruitment Details: College students seeking treatment at college counseling center. Eligible students endorsed suicidal thoughts at intake.
Pre-assignment Details: While they were consented to assure they fully understood the rights and responsibilities of their study role, data about Study Counselors is not collected as it is for the Student Participants. Per CT.gov request, they are however being included as a separate 8th Arm/Group for purposes of this data reporting.
Period: Overall Study
Arm/Group | CAMS to Maintenance | CAMS to CAMS | CAMS to DBT | TAU to Maintenance | TAU to CAMS | TAU to DBT | DBT Only | Study Counselors
Started | 12 | 8 | 10 | 4 | 7 | 1 | 26 | 16
Completed | 9 | 3 | 5 | 3 | 3 | 0 | 14 | 16
Not Completed | 3 | 5 | 5 | 1 | 4 | 1 | 12 | 0
Not completed — Lost to Follow-up | 3 | 0 | 0 | 1 | 1 | 0 | 2 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Treatment drop | 0 | 2 | 1 | 0 | 3 | 1 | 3 | 0
Not completed — Study drop | 0 | 3 | 3 | 0 | 0 | 0 | 7 | 0

BASELINE CHARACTERISTICS:
Population: While they were consented to assure they fully understood the rights and responsibilities of their study role, Study Counselors are not considered enrolled as study subjects. Therefore, they are not deemed a relevant Arm/group for reporting purposes here.
Groups:
- Total: Total of all reporting groups
Arm/Group | CAMS to Maintenance | CAMS to CAMS | CAMS to DBT | TAU to Maintenance | TAU to CAMS | TAU to DBT | DBT Only | Study Counselors | Total
Number analyzed (Participants) | 12 | 8 | 10 | 4 | 7 | 1 | 26 | 16 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] — {Note:While Counselor age data was provided, it was not included in determining the overall Mean and Standard deviations of the study participants because the study itself is focused on the students, including a maximum age Exclusion for student participants. Those numbers were derived for the 68 Student participants alone.}
  years | 21.08 (2.19) | 20.37 (2.07) | 20.90 (2.38) | 19.25 (1.26) | 19.86 (1.34) | 20.00 (8.00) | 19.88 (2.05) | 37.38 (9.05) | 20.26 (2.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 8 | 4 | 5 | 1 | 16 | 13 | 60
  Male | 4 | 3 | 2 | 0 | 2 | 0 | 10 | 3 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 6 | 8 | 3 | 5 | 1 | 17 | 1 | 50
  Not Hispanic or Latino | 3 | 2 | 2 | 1 | 2 | 0 | 9 | 15 | 34
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2
  Asian | 1 | 1 | 2 | 0 | 2 | 0 | 3 | 4 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Black or African American | 4 | 2 | 2 | 1 | 1 | 1 | 3 | 2 | 16
  White | 3 | 3 | 5 | 3 | 2 | 0 | 14 | 7 | 37
  More than one race | 3 | 1 | 1 | 0 | 0 | 0 | 4 | 2 | 11
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 8 | 10 | 4 | 7 | 1 | 26 | 16 | 84

OUTCOME MEASURES:

1. Primary Outcome: Number of Eligible Students Who Agree to Randomization
Description: Among students who are eligible to participate in the study and approached about the study by an intake worker, the number who agree to randomization to one of three treatments will be reported.
Time Frame: To the end of initial Randomization (up to 1 week)
Population: Students meeting all inclusion criteria and no exclusion criteria.
Measure: Count of Participants; unit: Participants
Groups:
- Duke University: Duke University (Durham, NC)
- Rutgers University: Rutgers University (New Brunswick, NJ)
- University of Nevada, Reno: University of Nevada, Reno
- University of Oregon: University of Oregon (Eugene, OR)
Arm/Group | Duke University | Rutgers University | University of Nevada, Reno | University of Oregon
Number analyzed (Participants) | 12 | 40 | 54 | 37
Participants | 8 | 24 | 20 | 16

2. Primary Outcome: Counselor Recruitment
Description: Among the counselors eligible to participate in the study, the number of counselors from each site who agree to participate.
Time Frame: To the end of initial counselor recruitment (up to 2 weeks)
Population: Counselors meeting all inclusion criteria and no exclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Duke University | Rutgers University | University of Nevada, Reno | University of Oregon
Number analyzed (Participants) | 4 | 4 | 4 | 4
Participants | 4 | 4 | 4 | 4

3. Primary Outcome: Treatment Adherence as Measured by DBT (Dialectical Behavior Therapy) Adherence Rating Scale
Description: Existing gold-standard adherence instruments for DBT will be used to rate a selection of sessions to assess counselors' fidelity to implementing the adaptive treatment strategies. Each item is rated on a scale where 0 = not used/not necessary, 1-3 = below adherence, 4 = minimum threshold for adherence, and 5 = adherent with high sufficiency. The DBT ACS is scored by averaging all non-zero items to create a computed global score where 3.8 and higher is considered "adherent."
Time Frame: To the end of treatment period (up to 16 weeks)
Population: Participants whose DBT sessions were rated.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Units Other Than Participants: sessions
Arm/Group | Duke University | Rutgers University | University of Nevada, Reno | University of Oregon
Number analyzed (Participants) | 2 | 4 | 4 | 4
Number analyzed (sessions) | 6 | 53 | 24 | 24
score on a scale | 3.5 [3.18 to 3.82] | 3.68 [3.61 to 3.75] | 3.72 [3.62 to 3.81] | 3.81 [3.74 to 3.89]

4. Primary Outcome: Treatment Adherence as Measured by CAMS (Collaborative Assessment and Management of Suicidality) Adherence Rating Scale
Description: Existing gold-standard adherence instruments for CAMS will be used to rate a selection of sessions to assess counselors' fidelity to implementing the adaptive treatment strategies. The measure consists of 14 items evaluating clinician performance, all rated on a seven-point Likert scale ranging from 0 ("Poor") to 6 ("Excellent"). A session is rated as adherent with a score of 3.5 or greater.
Time Frame: To the end of treatment period (up to 16 weeks)
Population: Participants whose CAMS sessions were rated.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Units Other Than Participants: sessions
Arm/Group | Duke University | Rutgers University | University of Nevada, Reno | University of Oregon
Number analyzed (Participants) | 2 | 4 | 3 | 4
Number analyzed (sessions) | 11 | 37 | 21 | 26
score on a scale | 4.05 [3.37 to 4.73] | 4.66 [4.32 to 5.01] | 4.45 [4.05 to 4.86] | 4.77 [4.39 to 5.15]

5. Primary Outcome: Number of Sessions Attended by Students in Each Treatment Condition
Time Frame: To the end of treatment period (up to 16 weeks)
Measure: Mean (Standard Deviation); unit: sessions
Arm/Group | CAMS to Maintenance | CAMS to CAMS | CAMS to DBT | TAU to Maintenance | TAU to CAMS | TAU to DBT | DBT Only
Number analyzed (Participants) | 12 | 8 | 10 | 4 | 7 | 1 | 26
sessions | 5.75 (1.14) | 5.75 (3.28) | 9.10 (3.41) | 6.00 (0.82) | 7.29 (3.35) | 7.00 (0.00) | 11.31 (4.54)

6. Primary Outcome: Number of Students Who Attrite From the Study (by Withdrawing Early From Treatment or Dropping Out of the Trial)
Time Frame: To the end of treatment period (up to 16 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | CAMS to Maintenance | CAMS to CAMS | CAMS to DBT | TAU to Maintenance | TAU to CAMS | TAU to DBT | DBT Only
Number analyzed (Participants) | 12 | 8 | 10 | 4 | 7 | 1 | 26
Participants | 0 | 5 | 4 | 0 | 3 | 1 | 10

7. Primary Outcome: Student Treatment Satisfaction as Measured by the Client Satisfaction Questionnaire (CSQ)
Description: CSQ items are rated from 1-4, with higher scores reflecting greater satisfaction.
Time Frame: To the end of treatment period (up to 16 weeks)
Population: Participants with data collected.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CAMS to Maintenance | CAMS to CAMS | CAMS to DBT | TAU to Maintenance | TAU to CAMS | TAU to DBT | DBT Only
Number analyzed (Participants) | 11 | 5 | 7 | 3 | 5 | 0 | 21
score on a scale
  Student CSQ at Stage 1 Treatment | 3.5 (0.42) | 3.4 (0.63) | 3.0 (0.73) | 3.83 (0.19) | 3.17 (0.57) |  | 3.31 (0.60)
  Student CSQ at Stage 2 Treatment: number analyzed (Participants) | 0 | 3 | 4 | 0 | 3 | 0 | 11
  Student CSQ at Stage 2 Treatment |  | 3.67 (0.38) | 2.47 (0.40) |  | 3.33 (0.52) |  | 3.63 (0.50)

8. Primary Outcome: Counselor Training Satisfaction
Description: An overall mean treatment satisfaction rating and the associated 95% confidence interval will be calculated based on counselors' responses on the Continuing Education Unit (CEU) evaluation surveys for the CAMS (Collaborative Assessment and Management of Suicidality) and DBT (Dialectical Behavior Therapy) online trainings. Item scores range from 1 (Not at all valuable) to 5 (Extremely valuable).
Time Frame: To end of initial training period (up to 4 weeks)
Population: We had 16 total consented counselors, and 2 entire rounds of DBT training, which some attended twice. 8 counselors attended both (8x2=16), while 4 others attended Round 1 only and another 4 attended Round 2 only. Therefore, a total of 24 DBT training ratings for 16 counselors. Ten counselors attended one CAMS session each.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Units Other Than Participants: Training sessions
Groups:
- Dialectical Behavior Therapy (DBT): Dialectical Behavior Therapy
- Collaborative Assessment and Management of Suicidality (CAMS): Collaborative Assessment and Management of Suicidality
Arm/Group | Dialectical Behavior Therapy (DBT) | Collaborative Assessment and Management of Suicidality (CAMS)
Number analyzed (Participants) | 16 | 10
Number analyzed (Training sessions) | 24 | 10
score on a scale | 4.48 [4.18 to 4.78] | 4.70 [4.40 to 5.00]

9. Primary Outcome: Counselor Assessment of Participant Study Satisfaction During Stage 1 of Treatment as Measured by the Client Satisfaction Questionnaire (CSQ)
Description: An overall mean treatment satisfaction rating and the associated 95% confidence interval will be calculated based on counselors' responses on the counselor version of the Client Satisfaction Questionnaire (CSQ). Items rated from 1-4, with higher scores reflecting greater satisfaction. Participants were assessed for overall mean treatment satisfaction rating based on counselors' responses on the counselor version of the Client Satisfaction Questionnaire (CSQ). The counselor version of the CSQ is completed by the counselor, based on their assessment of how the subject appreciated and benefited from treatment.
Time Frame: To the end of stage 1 (up to 8 weeks)
Population: Participants who completed Stage 1 of treatment.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | CAMS to Maintenance | CAMS to CAMS | CAMS to DBT | TAU to Maintenance | TAU to CAMS | TAU to DBT | DBT Only
Number analyzed (Participants) | 10 | 6 | 9 | 4 | 6 | 1 | 24
score on a scale | 3.46 [3.32 to 3.60] | 2.96 [2.71 to 3.21] | 2.92 [2.68 to 3.16] | 3.56 [3.37 to 3.75] | 2.79 [2.70 to 2.88] | 2.88 [2.88 to 2.88] | 2.96 [2.85 to 3.07]

10. Primary Outcome: Counselor Assessment of Participant Study Satisfaction During Stage 2 of Treatment as Measured by the Client Satisfaction Questionnaire (CSQ)
Description: as for outcome 9
Time Frame: Beginning to end of Stage 2 (up to 8 weeks)
Population: Participants who completed Stage 2 of treatment.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | CAMS to Maintenance | CAMS to CAMS | CAMS to DBT | TAU to Maintenance | TAU to CAMS | TAU to DBT | DBT Only
Number analyzed (Participants) | 0 | 3 | 6 | 0 | 4 | 0 | 18
score on a scale |  | 2.88 [2.75 to 3.01] | 2.90 [2.68 to 3.12] |  | 3.00 [3.00 to 3.00] |  | 3.24 [3.08 to 3.40]

ADVERSE EVENTS:
Time Frame: To the end of study (up to 9 months)
Description: While consented to assure they fully understood the rights and responsibilities of their study role, Study Counselors are not considered enrolled as study subjects. They are not deemed a relevant Arm/group for reporting purposes here. Adverse Events were only collected in regards to treatment subjects.
  Regarding Arm "DBT Only", there was no formal separation into Stage 1/2 of treatment as it was one, longer, course of DBT. Therefore, all related data is accumulated under that single Arm.
Groups:
- Stage 2 - CAMS to Maintenance: Subject assigned to CAMS for Phase 1. Subject is a Phase 1 CAMS Responder, thus placed into ongoing Maintenance/Monitoring.
  CAMS - Phase 1: 4-8 weeks of CAMS treatment
- Stage 2 - CAMS to CAMS: Subject assigned to CAMS for Phase 1. Subject is a Phase 1 CAMS Insufficient Responder, then assigned to Phase 2 CAMS.
  CAMS - Phase 1: 4-8 weeks of CAMS treatment
  CAMS - Phase 2: Up to 8 weeks of CAMS treatment
- Stage 2 - CAMS to DBT: Subject assigned to CAMS for Phase 1. Subject is a Phase 1 CAMS Insufficient Responder, then assigned to Phase 2 DBT.
  CAMS - Phase 1: 4-8 weeks of CAMS treatment
  DBT - Phase 2: Up to 8 weeks of DBT treatment
- Stage 2 - TAU to Maintenance: Subject assigned to TAU for Phase 1. Subject is a Phase 1 TAU Responder, thus placed into ongoing Maintenance/Monitoring.
  TAU - Phase 1: 4-8 weeks of TAU treatment
- Stage 2 - TAU to CAMS: Subject assigned to TAU for Phase 1. Subject is a Phase 1 TAU Insufficient Responder, then assigned to Phase 2 CAMS.
  TAU - Phase 1: 4-8 weeks of TAU treatment
  CAMS - Phase 2: Up to 8 weeks of CAMS treatment
- Stage 2 - TAU to DBT: Subject assigned to TAU for Phase 1. Subject is a Phase 1 TAU Insufficient Responder, then assigned to Phase 2 DBT.
  TAU - Phase 1: 4-8 weeks of TAU treatment
  DBT - Phase 2: Up to 8 weeks of DBT treatment
- DBT Only: Subject Assigned to DBT for Phase 1, continuing up to 16 weeks.
  No 2nd phase is delineated.
- Stage 1 CAMS: All Subjects assigned to Stage 1 CAMS who had a relevant AE during Stage 1.
- Stage 1 TAU: All Subjects assigned to Stage 1 TAU who had a relevant AE during Stage 1.
Arm/Group | Stage 2 - CAMS to Maintenance | Stage 2 - CAMS to CAMS | Stage 2 - CAMS to DBT | Stage 2 - TAU to Maintenance | Stage 2 - TAU to CAMS | Stage 2 - TAU to DBT | DBT Only | Stage 1 CAMS | Stage 1 TAU
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/5 | 0/9 | 0/4 | 0/7 | 0/1 | 0/26 | 0/30 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/8 | 0/9 | 0/4 | 0/7 | 0/1 | 4/26 | 4/30 | 1/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/5 | 1/9 | 0/4 | 0/7 | 0/1 | 3/26 | 9/30 | 3/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Stage 2 - CAMS to Maintenance (N=12) | Stage 2 - CAMS to CAMS (N=8) | Stage 2 - CAMS to DBT (N=9) | Stage 2 - TAU to Maintenance (N=4) | Stage 2 - TAU to CAMS (N=7) | Stage 2 - TAU to DBT (N=1) | DBT Only (N=26) | Stage 1 CAMS (N=30) | Stage 1 TAU (N=12)
Suicide Attempt (Psychiatric disorders) | 0 | 0/5 | 0 | 0 | 0 | 0 | 1 | 3 | 1
Suicidal Ideation (Psychiatric disorders) | 0 | 0/5 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Non-suicidal self-injury (Psychiatric disorders) | 0 | 0/5 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Other non-mental health event (General disorders) | 0 | 0/5 | 0 | 0 | 0 | 0 | 2 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stage 2 - CAMS to Maintenance (N=12) | Stage 2 - CAMS to CAMS (N=5) | Stage 2 - CAMS to DBT (N=9) | Stage 2 - TAU to Maintenance (N=4) | Stage 2 - TAU to CAMS (N=7) | Stage 2 - TAU to DBT (N=1) | DBT Only (N=26) | Stage 1 CAMS (N=30) | Stage 1 TAU (N=12)
Evidence of distress during assessments (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 9 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-04-08): https://cdn.clinicaltrials.gov/large-docs/15/NCT04728815/Prot_SAP_001.pdf
  • Informed Consent Form (2022-03-31): https://cdn.clinicaltrials.gov/large-docs/15/NCT04728815/ICF_000.pdf